CLINICAL TRIAL: NCT01768260
Title: Study of the Effect of EECP on Anterior Ischemic Optic Neuropathy
Brief Title: Effect of EECP on Anterior Ischemic Optic Neuropathy
Acronym: AION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, WenHui Zhu, Oculist-in-charge, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eye EECP-1
Record Dates: First submitted 2013-01-08; First posted 2013-01-15 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Anterior Ischemic Optic Neuropathy
Keywords: visual acuity; artery flow velocity; Enhanced External Counterpulsation; Ischemic; Optic Neuropathy
MeSH Terms: conditions — Optic Neuropathy, Ischemic; Ischemia; Optic Nerve Diseases | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced External conterpulsation (Active Comparator): Enhanced external counterpulsation (EECP) is a noninvasive modality for the treatment of ischemic cardiovascular disease. EECP therapy is done by sequential inflation of 3 sets of cuffs wrapped around the lower extremities during diastole and deflation of the cuffs during systole.
  Interventions: Device: Enhanced external counterpulsation; Drug: Aspirin
- aspirin (Active Comparator): The subjects with Anterior ischemic Optic Neuropathy received aspirin therapy.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Device: Enhanced external counterpulsation — EECP is performed for 1 hours every day, for a total of 36 hours.
  Other Names: EECP
  Arms: Enhanced External conterpulsation
Drug: Aspirin — Standard drug therapy

SUMMARY:
Enhanced External Counterpulsation(EECP) therapy may promote the recovery of visual function by improving the blood perfusion of eyes. The present study aims to investigate the effect of EECP on Anterior Ischemic Optic Neuropathy.

DETAILED DESCRIPTION:
Patients with Anterior Ischemic Optic Neuropathy are randomized into two groups: one group receive standard medical treatment for ischemic optic neuropathy, the other group plus EECP therapy besides standard medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* ischemic optic neuropathy
* within 1 month

Exclusion Criteria:

* Hemorrhagic disease
* thrombophlebitis or infection lesions
* severe hypertensive patients
* Atrial fibrillation
* Aortic regurgitation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
visual acuity | 7 weeks

SECONDARY OUTCOMES:
Ophthalmic artery blood flow velocity | 7 weeks

OTHER OUTCOMES:
Central retinal artery flow velocity | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yan Zhang, Professor, Study Director — First Affiliated Hospital of Sun Yat-sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat- sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Werner D, Michalk F, Harazny J, Hugo C, Daniel WG, Michelson G. Accelerated reperfusion of poorly perfused retinal areas in central retinal artery occlusion and branch retinal artery occlusion after a short treatment with enhanced external counterpulsation. Retina. 2004 Aug;24(4):541-7. doi: 10.1097/00006982-200408000-00006. PMID 15300074